Study of the Efficacy of GGED: a Cognitive Training App for Eating Disorders.

NCT06179992 22/12/2023

## STATISTICAL ANALYSIS PLAN

Descriptive statistics will be used to report means, standard deviances and frequencies. In addition, tests will be performed to evaluate differences between the different variables considered in the study. To predict the different response variables under study, generalised linear mixed model (GLMM) will be carried out. Specifically, a multiple linear regression model, where the outcomes measures are dependant variables, whereas the independent variable is time: T1, T2, T3.